CLINICAL TRIAL: NCT03129737
Title: Multi-centre Randomised Trial Investigating the Effect of PROphylactic triCuspID Annuloplasty in Patients With Dilated Tricuspid Annulus on Tricuspid Regurgitation Progression, Right Ventricular Remodeling and Functional Outcomes
Brief Title: PROphylactic triCuspID Annuloplasty in Patients With Dilated Tricuspid Annulus
Acronym: PROCIDA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ettore Sansavini Health Science Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ESREFO 18
Record Dates: First submitted 2017-04-18; First posted 2017-04-26 (Actual); Last update posted 2017-06-28 (Actual); Status verified 2017-06

CONDITIONS: Tricuspid (Valve) Insufficiency (Rheumatic)
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tricuspid valve annuloplasty (Experimental): Concomitant tricuspid valve annuloplasty in patients with tricuspid annulus dilatation (>21mm /m2) with or without TR≤ moderate in pts undergoing mitral valve surgery
  Interventions: Procedure: Mitral valve surgery; Procedure: Tricuspid valve annuloplasty
- Mitral valve repair (Active Comparator): No concomitant tricuspid valve annuloplasty in patients with tricuspid annulus dilatation (>21mm/m2) with or without TR ≤ moderate in pts undergoing mitral valve surgery
  Interventions: Procedure: Mitral valve surgery

INTERVENTIONS:
Procedure: Mitral valve surgery — Mitral valve repair is preferred whenever technically feasible over valve replacement. Annuloplasty may be used as sole therapy or in conjunction with other repair maneuvers to support the reconstruction and reinforce the annulus as well as prevent future annular dilatation. The mitral regurgitation secondary to myxomatous degeneration is prolapse of the middle scallop of the posterior leaflet result from chordal rupture or chordal elongation. Quadrangular resection of the involved middle scallop of the posterior leaflet combined with a posterior mitral annuloplasty is the best way to handle this situation. Chordae replacement could be used also to treat flail/prolapse of the anterior leaflet. Annuloplasty is always doing in mitral valve repair to stabilize and reshape the annulus.
Procedure: Tricuspid valve annuloplasty — Depending on the extent of the valve disease, there is the possibility to perform valve repair. In mitral valve reference center the rate of repair will reach 100%. In many patients with mitral valve regurgitation, tricuspid valve will be insufficient or the annulus dilated. Tricuspid annuloplasty ring will be helpful to treat dilation by reshaping, or to treat the regurgitant diseases. The ring will be secured and sutured to the native annulus by U-stitches.
  Arms: Tricuspid valve annuloplasty

SUMMARY:
Patients elected to undergo mitral valve surgery (either repair or replacement) with less equal than moderate (≤+2) tricuspid regurgitation and dilated tricuspid annulus (>21mm/m2) at preoperative echocardiography will be screened. Consenting patients fulfilling all inclusion and exclusion criteria will be included in the study and assigned to elective mitral valve replacement or repair with or without concomitant tricuspid annuloplasty in a 1:1 fashion, using a blocked randomization scheme balanced within center.

DETAILED DESCRIPTION:
The present study is designed as a prospective, multicentre, multinational, randomized, 2-arm parallel group trial. Participating centres are selected based on previous experience with the surgical technique and standardised echo imaging. Each center is expected to contribute 20 to 40 patients over a 12-month enrolment period.

Patients elected to undergo mitral valve surgery (either repair or replacement) with less equal than moderate (≤+2) tricuspid regurgitation and dilated tricuspid annulus (>21mm/m2) at preoperative echocardiography will be screened. Consenting patients fulfilling all inclusion and exclusion criteria will be included in the study and assigned to elective mitral valve replacement or repair with or without concomitant tricuspid annuloplasty in a 1:1 fashion, using a blocked randomization scheme balanced within center.

After discharge patients will be assessed at 1 month (phone contact), 6 month and 1-year after surgery.

ELIGIBILITY:
Inclusion Criteria:

Patients undergoing mitral valve surgery (either repair or replacement) with less/equal than moderate (≤+2) tricuspid regurgitation and dilated tricuspid annulus (>21mm/m2 BSA) at preoperative echocardiography and fulfilling the following selection criteria:

Inclusion criteria:

1. Written informed consent
2. Degenerative mitral valve disease
3. > 18 years old

Exclusion Criteria:

Main exclusion criteria:

1. Presence of structural or organic tricuspid valve disease
2. urgent operation
3. presence of pacemaker leads through the tricuspid annulus
4. acute endocarditis or other organic valve diseases
5. previous surgical procedure
6. Severe TR
7. Associated cardiac procedure
8. NYHA class IV
9. Severe COPD (GOLD class 3,4)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-05-17 (Actual); Primary Completion 2020-02 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Progression of TR | 1 year
  Progression of TR at one year follow-up defined as worsening of at least one class with respect to pre-surgery as assessed by the Core lab evaluation of the echocardiogram.

SECONDARY OUTCOMES:
Evaluation of reverse right ventricle (RV) remodelling | 1 year
  The evaluation of reverse right ventricle (RV) remodelling, assessed as reduction/modification of the end diastolic and end systolic RV diameters with respect to pre-surgery
Residual TR | 1 year
  Percentage of patients with moderate to severe TR at one year after surgery

OTHER OUTCOMES:
NYHA Class | 1 year
  Modification of NYHA class at one year after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Maria Salomone, MD, Study Director — Fondazione Ettore Sansavini per la Ricerca Scientifica ONLUS
Locations (8):
- Italy (8):
  - Casa di Cura Montevergine, Mercogliano, Avellino
  - ICLAS, Rapallo, Genova
  - Maria Cecilia Hospital, Cotignola, Ravenna
  - Anthea Hospital, Bari
  - Ospedale Santa Maria, Bari
  - Città di Lecce Hospital, Lecce
  - Maria Eleonora Hospital, Palermo
  - Maria Pia Hospital, Torino

IPD SHARING:
Plan to Share IPD: No